CLINICAL TRIAL: NCT02940132
Title: Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics/ Pharmacodynamics and Preliminary Efficacy of SC10914 in Patients With Advanced Solid Tumors
Brief Title: A Study of SC10914 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QF-SC10914-011
Record Dates: First submitted 2016-10-08; First posted 2016-10-20 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2016-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SC10914 (Experimental): SC10914 Dose Escalation： Dose Level 1：30mg(QD) Dose Level 2：60mg(QD) Dose Level 3：120mg(QD) Dose Level 4：200mg(QD) Dose Level 5：100mg(BID) Dose Level 6：300mg(QD) Dose Level 7：150mg(BID) Dose Level 8：400mg(QD) Dose Level 9：200mg(BID) Dose Expansion： Receiving SC10914 in one of three dosage regimens(low, middle or high dose-level and QD or BID) based on the assessment of dose escalation study.
  Interventions: Drug: SC10914

INTERVENTIONS:
Drug: SC10914 — SC10914 will be administered orally.

SUMMARY:
SC10914 is a potent selective PARP-1 and PARP-2 inhibitor. This study aims to determine the safety , tolerability , pharmacokinetic/pharmacodynamics profile of increasing doses of SC10914 when administered orally to patients with advanced solid tumors. Furthermore, the safety and efficacy of SC10914 in patients with advanced solid tumors and negative expression of ATM or BRCA1 or BRCA2 mutation will be evaluated in expanded cohorts to establish the Recommended Phase 2 Dose(RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged 18-70 years
* Dose escalation study: Subjects diagnosed with advanced solid malignancies who are refractory to standard therapies or for which no standard therapy exists/Dose Expansion study: Subjects diagnosed with advanced solid malignancies who are refractory to standard therapies or for which no standard therapy exists and negative expression of ATM or BRCA1 or BRCA2 mutation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Have measurable lesion exists(RECIST 1.1)
* Life expectancy≥3 months
* Have adequate bone marrow, hepatic and renal functions

Exclusion Criteria:

* Allergic constitution or hypersensitivity to investigational drugs or relevant drug
* Patients who received any previous treatment with a PARP inhibitor
* Patients accepted anti-cancer therapy including chemotherapy, radiotherapy, endocrinotherapy, immunotherapy, Chinese herbal treatment or other investigational drugs within 4 weeks prior to trial entry (or a longer period depending on the defined characteristics of the drugs used eg,. 6 weeks for mitomycin C or nitrosourea)
* With serious pre-existing medical conditions, such as significant cardiovascular disease and psychogenic disorders
* With family history of long QT syndrome or QTc ≥ 450 ms
* With persistent CTCAE ≧grade 2 toxicities (excluding alopecia) caused by prior medication
* With symptomatic brain metastases
* Pregnancy or lactation
* With Hepatitis B or C or human immunodeficiency virus infections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Study: Maximum-tolerated Dose (MTD) of SC10914 | 30 days
  In dose escalation study, SC10914 will be administered to patients with advanced solid tumors. MTD is defined as the maximum dose level at which no more than one subject out of three experiences has a dose-limiting toxicity (DLT) within 30 days after accepting SC10914.
Dose Expansion Study: Recommended Phase II Dose(RP2D) of SC10914 | 8 weeks
  In dose expansion study,SC10914 will be administered to patients with advanced solid tumors and negative expression of ATM or BRCA1 or BRCA2 mutation.RP2D will be defined based on all available safety, pharmacokinetics(PK), pharmacodynamics(PD), and efficacy data collected after the start of SC10914 treatment.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) as assessed by NCI-CTCAE v4.03 | 8 weeks
Area under the concentration-time curve (AUC) | 4 weeks
Time to reach maximum concentration (Tmax) | 4 weeks
Maximum Concentration (Cmax) | 4 weeks
Trough Concentration (Ctrough) | 4 weeks
Elimination Half-Life (T½) | 4 weeks
Clearance (CL) | 4 weeks
Volume of Distribution (Vd) | 4 weeks
Evaluation of the effects of PARP inhibition of SC10914 by the peripheral blood mononuclear cells（PBMC） | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by overall response rate (ORR) | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by disease control rate (DCR) | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by progression free survival (PFS) | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by duration of response (DOR) | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by time to progression (TTP) | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by overall survival (OS) | Baseline until death
Evaluation of the antitumor effects of SC10914 as measured by tumor markers CA-125 as assessed by Gynecologic Cancer Intergroup(GCIG) | 8 weeks
Evaluation of the antitumor effects of SC10914 as measured by tumor markers PSA as assessed by Prostate-Specific Antigen Working Group(PSAWG) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes